CLINICAL TRIAL: NCT01537354
Title: A Comparison of Immediate Changes in Pulmonary Compliance Between Curosurf and Survanta in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Comparison in Pulmonary Compliance Between Curosurf and Survanta in Preterm Infants With Respiratory Distress Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discontinued clinical trial before enrollment of subjects.
Sponsor: University of Michigan (Other)
Collaborators: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Steven Donn, M.D., Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Curosurf-Survanta-UM13888
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — poractant alfa; beractant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Survanta® (Active Comparator): Survanta® (Beractant, Abbot Laboratories, Columbus, OH) Surfactant will be administered by respiratory therapist not involved in patient's care.
  Interventions: Drug: Survanta®
- Curosurf® (Active Comparator): Curosurf® (Cornerstone Therapeutics, Inc., Cary, NC Surfactant will be administered by respiratory therapist not involved in patient's care.
  Interventions: Drug: Curosurf®

INTERVENTIONS:
Drug: Curosurf® — Initial dose is 2.5ml/kg (200 mg/kg phospholipid) administered via endotracheal tube. Subsequent doses if needed are 1.25 mL/kg (100 mg/kg phospholipids).
  Arms: Curosurf®
Drug: Survanta® — Initial dose is 4 mL/kg (100 mg/kg phospholipids) administered via endotracheal tube. Subsequent doses if needed are 4 mL/kg (100 mg/kg phospholipids).
  Arms: Survanta®

SUMMARY:
This is a null hypothesis study. The investigators hypothesize that there will be no difference in changes in dynamic compliance when measured at 15, 30, 45 and 60 minute intervals after administration of either surfactant and there will be no differences in the number of doses needed between the two surfactants in premature infants admitted to our NICU.

DETAILED DESCRIPTION:
Premature newborn infants may have impaired lung function as a result of their prematurity. When this occurs, the newborns show poor oxygen and carbon dioxide exchange and difficulty in breathing. The reason for these symptoms is due in part to the lack of special chemicals in the lungs, called phospholipids or surfactant. The lack of these special chemicals causes the babies lung to be difficult to ventilate. Treatment of this condition can require placing an artificial airway (endotracheal tube) into the babies windpipe (intubation) and use of a breathing machine (ventilator). In addition, physicians frequently give these special chemicals (phospholipid) through the childs airway. There are several different types of phospholipids available for this treatment in newborns but very limited amount of studies have been done to examine differences in the ability to ventilate between the various types of surfactant. The investigators propose to examine immediate changes in ability to ventilate (dynamic compliance) at specific time intervals after administration of either type of surfactant; Curosurf or Survanta.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 28 and 31 6/7 weeks' gestational age
* Inborn to UM NICU
* < 12 hours of age
* Respiratory Distress Syndrome
* radiographic evidence
* need for endotracheal intubation
* Oxygen requirement > 30% FiO2
* Decision to give surfactant by the treatment team

Exclusion Criteria:

* Major congenital anomaly
* Sepsis syndrome in extremis

Ages: 15 Minutes to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in dynamic compliance | 15 minutes, 30 minutes, 45 minutes and then hourly intervals after administration of surfactant. Subjects' compliance will be monitored hourly after the first 60 minutes while they are being ventilated in the Neonatal Intensive Care Unit.
  Patient's dynamic compliance will be measured immediately after initial dosage, q15 minutes for 60 minutes and hourly for 48 hrs as long as intubated.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Donn, M.D., Principal Investigator — University of Michigan C & W Mott Children's Hospital
Locations (1):
- University of Michigan C & W Mott Children's Hospital, Ann Arbor, Michigan, United States